CLINICAL TRIAL: NCT02635997
Title: Antiresorptive Effects of a 6-m Treatment Course With Ibandronate Plus Supplementation of Vitamine D and Calcium in Central America
Status: Completed | Type: Observational
Sponsor: Pontifical Catholic University of Argentina (Other)
Responsible Party: Principal Investigator, Santiago Perez Lloret, Associate Researcher, Pontifical Catholic University of Argentina
Other Study IDs: Catholic University
Record Dates: First submitted 2015-12-13; First posted 2015-12-21 (Estimated); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Osteoporosis
Keywords: osteoporosis; ibandronate; vitamine D; calcium; bone mineral density; health-related quality of life
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients on antiresorptive therapy: Ibandronate 150 mg per month + Vitamine D 400-800 IU and Calcium 500-1000 mg per day
  Interventions: Drug: antiresorptive therapy

INTERVENTIONS:
Drug: antiresorptive therapy

SUMMARY:
Ibandronate is a third-generation biphosphonate with recognized antiresorptive efficacy by several international, randomized, double-blind, controlled trials. These studies have not included patients from central america, to the best of our knowledge. Therefore, this open-label, uncontrolled study, was set out to assess the clinical effects of a 6-m treatment course with Ibandronate plus vitamine D and Calcium on bone mineral density and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women with a diagnosis of osteoporosis of at-Risk
* Have a medical indication to receive Ibandronate+Vitamine D+Calcium

Exclusion Criteria:

* Osteoporosis due to secondary causes

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with a diagnosis of osteoporosis o with a high risk of developing it in the near future.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | 6 months
Health-Related Quality of Life | 6 months

SECONDARY OUTCOMES:
Adverse Events | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University, Buenos Aires, Argentina